CLINICAL TRIAL: NCT00112632
Title: Open-Label Trial of Neoadjuvant Imatinib Mesylate (Glivec) in Patients With Locally Advanced Malignant Gastrointestinal Stromal Tumors (GIST) Expressing c-Kit or Platelet-Derived Growth Factor Receptor-alpha
Brief Title: Imatinib Mesylate in Treating Patients With Locally Advanced Gastrointestinal Stromal Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000430499; KRDI-TUM-GIST-CST1571-BDE43; EU-20507
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: gastrointestinal stromal tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate; Neoadjuvant Therapy

INTERVENTIONS:
Drug: imatinib mesylate
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving imatinib mesylate before surgery may shrink the tumor so that it can be removed.

PURPOSE: This phase II trial is studying how well imatinib mesylate works in treating patients with locally advanced gastrointestinal stromal tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine radiographic objective response rates in patients with locally advanced gastrointestinal stromal tumor treated with neoadjuvant imatinib mesylate.
* Determine histological response in patients treated with this drug.

Secondary

* Determine R0-resectability and organ-preserving resectability in these patients after treatment with this drug.
* Correlate radiographic imaging and metabolic imaging with histological response in patients treated with this drug.
* Determine the safety and tolerability of this drug in these patients.

OUTLINE: This is a nonrandomized, open-label, multicenter study.

Patients receive oral imatinib mesylate once or twice daily for 4-6 months in the absence of disease progression or unacceptable toxicity. Within 2-3 weeks after completion of imatinib mesylate, patients with responding or stable disease undergo surgical resection.

After completion of study treatment, patients are followed at 4 weeks, 6 months, and then at 1 year.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed gastrointestinal stromal tumor

  * Locally advanced disease
  * Potentially resectable disease*

    * No tumor that can be completely resected (R0) with sufficient margins NOTE: *Multivisceral resection may be necessary
* Tumor must stain positive for c-Kit (CD117) or platelet-derived growth factor receptor-alpha (PDGFRA) by immunohistochemistry
* At least 1 site of measurable disease
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-3

Life expectancy

* Not specified

Hematopoietic

* Platelet count > 100,000/mm^3
* Absolute neutrophil count > 1,500/mm^3

Hepatic

* AST and ALT < 2.5 times upper limits of normal (ULN) (5 times ULN if hepatic metastases are present)
* Bilirubin < 1.5 times ULN
* No chronic active hepatitis
* No cirrhosis
* No other chronic liver disease

Renal

* Creatinine < 1.5 times ULN
* No chronic renal disease

Cardiovascular

* No New York Heart Association class III-IV cardiac disease
* No congestive heart failure
* No myocardial infarction within the past 6 months

Immunology

* No active uncontrolled infection
* No known HIV positivity

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after completion of study treatment
* Must be medically fit to undergo surgery
* No other primary malignancy within the past 5 years except basal cell skin cancer, carcinoma in situ of the cervix, or a primary malignancy that is not currently clinically significant and does not require active intervention
* No gastrointestinal obstruction or major bleeding episode requiring immediate surgical intervention
* No uncontrolled diabetes
* No other severe or uncontrolled medical disease
* No significant history of noncompliance to medical regimens

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent anticancer biologic agents

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosourea or mitomycin) unless disease is rapidly progressing
* No concurrent anticancer chemotherapy

Endocrine therapy

* No concurrent systemic corticosteroid therapy unless approved by the study sponsor

Radiotherapy

* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to ≥ 25% of bone marrow

Surgery

* More than 2 weeks since prior major surgery except tumor biopsy

Other

* More than 4 weeks since prior investigational drugs unless disease is rapidly progressing
* No other concurrent anticancer therapy
* No other concurrent investigational agents
* No concurrent warfarin for therapeutic anticoagulation

  * Concurrent low molecular weight heparin (e.g., enoxaparin sodium) or heparin for therapeutic anticoagulation allowed
  * Concurrent mini-dose warfarin (e.g.,1 mg/day) for prophylaxis of central venous catheter thrombosis allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-02

PRIMARY OUTCOMES:
Overall tumor response (complete response, partial response, stable disease, and progression of disease)

SECONDARY OUTCOMES:
Time to progression of disease
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Licht, MD, Study Chair — Technical University of Munich
Locations (9):
- Allgemeines Krankenhaus - Universitatskliniken, Vienna, Austria
- Germany (8):
  - Robert Roessle Comprehensive Cancer Center - Charite Campus Buch, Berlin
  - Universitaetsklinikum Bonn, Bonn
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - University Medical Center Hamburg - Eppendorf, Hamburg
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Southwest German Cancer Center at Eberhard-Karls-University, Tübingen
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden